CLINICAL TRIAL: NCT02219152
Title: Topical Instillation of Tranexamic Aacid in Bronchoscopy to Decrease Bleeding During Entobronchial & Transbronchial Biopsiy: a Prospective Double Blind Placebo Controlled Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liran Levy (Other)
Responsible Party: Sponsor-Investigator, Liran Levy, Topical Instillation of Tranexamic Aacid in Bronchoscopy to Decrease Bleeding During Entobronchial & Transbronchial Biopsiy: a Prospective Double Blind Placebo Controlled Study, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0321-14
Record Dates: First submitted 2014-08-12; First posted 2014-08-18 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Bronchoscopy Biopsy
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tranexamic acid (Experimental): tranexamic acid will be administrated using the bronchoscope
  Interventions: Drug: tranexamic acid
- saline (Placebo Comparator): the saline will be administrated using an infusion during the biopsy.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: tranexamic acid
  Arms: tranexamic acid
Drug: saline
  Arms: saline

SUMMARY:
Bleeding during transbronchial ro endobronchial biopsy is rather a common complication.

Mostly this is an insignificant bleeding, but in 3% of the biopsies there is a substantial amount of bleeding that requires a special treatment or follow up.

The goal of this study is to examine whether submission of tranexamic acid during the biopsy could diminish the amount of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patient that are candidates to endobronchial or transcronchial biopsy

Exclusion Criteria:

* S/P MI or CVA or PE or DVT .
* S/P thrombophilia.
* Patients under coagulation therpay
* Chronic Renal Failure
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
amount of bleeding | participants will be followed for the duration of hospital stay, an expected average of one day
  amount of bleedibg that will be calculated on the basis of the difference between the amount of saline that will be injected at the bronchoscopy and the blood and fluid that will be collected in the suction tank.

SECONDARY OUTCOMES:
amount of erythrocytes | participants will be followed for the duration of hospital stay, an expected average of one day
  amount of erythrocytes by multiplying the Hematocrit and blood volume

CONTACTS AND LOCATIONS:
Overall Officials: Neville Berkman, MD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel